CLINICAL TRIAL: NCT02382016
Title: A Randomized, Double-blind, Placebo-controlled, Prospective, Multicenter, Parallel Group Study to Assess the Safety and Efficacy of Macitentan in Patients With Portopulmonary Hypertension
Brief Title: PORtopulmonary Hypertension Treatment wIth maCitentan - a randOmized Clinical Trial
Acronym: PORTICO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055-404
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Portopulmonary Hypertension
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational treatment (Experimental): Macitentan film-coated tablet 10 mg once daily.
  Interventions: Drug: Macitentan
- Placebo (Placebo Comparator): Matching placebo tablet once daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Macitentan — Macitentan film-coated tablet 10 mg once daily.
  Other Names: ACT-064992
  Arms: Investigational treatment
Other: Placebo — Matching placebo tablet once daily.
  Arms: Placebo

SUMMARY:
24-week study to evaluate the efficacy and safety of macitentan for the treatment of portopulmonary hypertension.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female of at least 18 years of age
* Confirmed diagnosis of portopulmonary hypertension

Main Exclusion Criteria:

* Severe hepatic impairment
* Severe obstructive or restrictive lung disease
* Pulmonary veno-occlusive disease
* Systolic blood pressure (SBP) < 90 mmHg at Screening
* ALT/AST >= 3 x ULN
* Bilirubin >= 3 mg/dL at Screening
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Perchenet, PhD, Study Director — Actelion
Locations (52):
- United States (29):
  - Mayo Clinic -Clinical Studies Unit, Phoenix, Arizona
  - UCSD, La Jolla, California
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - Keck School of Medicine, Los Angeles, California
  - UCSF, San Francisco, California
  - University of Colorado Health Sciences Center Aurora, Aurora, Colorado
  - University of Florida - Divison of Pulmonary Critical Care & Sleep, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Mayo Clinic Florida - Pulmonary Dept., Jacksonville, Florida
  - University of Miami, Miami, Florida
  - South Miami Hospital, South Miami, Florida
  - Emory Healthcare, Atlanta, Georgia
  - Piedmont Healthcare, Austell, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Boston University, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic - Department of Cardiovascular Medicine, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Montefiore, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center Division of NeuroCritical Care 75390-8550, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin
- Brazil (2):
  - Servico de Hipertensao Pulmonar - Complexo Hospitalar Santa Casa Irmandade Santa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo (HC-FMUSP), São Paulo
- Czechia (2):
  - Lékařská fakulta a Všeobecná fakultní nemocnice v Praze, II. Interní klinika kardiologie a angiologie U, Prague
  - IKEM (Institut klinické a experimentální medicíny, Institute for Clinical and Experimental Medicine), Prague
- France (9):
  - CHRU de Grenoble, Hôpital Albert Michallon, Grenoble, Auvergne-Rhône-Alpes
  - CHRU Hôpital Cavale Blanche Brest, Brest, Brittany Region
  - CHU Côte de Nacre, Service de Pneumologie, Caen
  - Hôpital cardiologique, Service de cardiologie 59037 Lille Cedex", Lille
  - Hôpital Cardiologique et Pneumologique Louis Pradel 69677 Bron cedex", Lyon
  - Hôpital Kremlin Bicêtre Service de Pneumologie, Paris
  - Hôpital Pontchaillou - CHU Rennes Service de Cardiologie et des Maladies Vasculaires Rennes Cedex 9 35033", Rennes
  - CHU Rouen, Rouen
  - CHU Toulouse - Hôpital Larrey Hôpital de Jour et Semaine, Toulouse
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Giessen und Marburg GmbH Justus-Liebig Universität Giessen 35392, Giessen
  - Medizinische Hochschule Hannover, Abteilung Pneumologie, Hanover
  - Thoraxklinik des Universitätsklinikums Heidelberg Zentrum für pulmonale Hypertonie Studienkoordination, Heidelberg
  - Universitätsklinikum Leipzig, Department Innere Medizin, Abteilung Pneumologie, Leipzig
- Spain (2):
  - Hospital Clinico i Provincial Servicio de Neumología, Barcelona
  - Hospital Universitario12 Octubre, Madrid
- United Kingdom (3):
  - NHS Greater Glasgow and Clyde Trust, Glasgow, Scotland
  - The Royal Free Hospital/ Cardiology Department, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Raevens S, Fallon MB. PORTICO: First Randomized Controlled Trial of Vasomodulator Therapy in Portopulmonary Hypertension. Hepatology. 2020 May;71(5):1870-1872. doi: 10.1002/hep.31166. No abstract available. PMID 32031690
- [Derived] Sitbon O, Bosch J, Cottreel E, Csonka D, de Groote P, Hoeper MM, Kim NH, Martin N, Savale L, Krowka M. Macitentan for the treatment of portopulmonary hypertension (PORTICO): a multicentre, randomised, double-blind, placebo-controlled, phase 4 trial. Lancet Respir Med. 2019 Jul;7(7):594-604. doi: 10.1016/S2213-2600(19)30091-8. Epub 2019 Jun 6. PMID 31178422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at 39 sites in 7 countries were screened and were randomized at 36 sites in these 7 countries (Brazil, Czech Republic, France, Germany, Spain, UK and US).
Pre-assignment Details: A total of 119 participants were screened and 85 participants were randomized (43 to macitentan 10 mg once daily and 42 to matching placebo) and received double-blind (DB) study treatment. Overall, 80 participants who completed DB treatment period entered the open-label (OL) treatment period and 33 participants in open-label extension (OLE) period.
Groups:
- Macitentan 10 mg: Participants received Macitentan 10 milligram (mg) film-coated tablets orally once daily for 12 weeks in Double-blind treatment period. Participants who completed DB treatment period continued to receive macitentan 10 mg for 12 weeks (up to Week 24) in OL treatment period . Participants (who were randomized at French sites) who completed the core phase of the study as scheduled and opted to continue receiving OL study treatment continued to receive macitentan 10 mg in OLE period.
- Placebo: Participants received Macitentan matching placebo film-coated tablets orally once daily for 12 weeks in Double-blind treatment period. Participants who completed DB treatment period were administered with macitentan 10 mg for 12 weeks (up to Week 24) in OL treatment period. Participants who were randomized at French sites who completed the core study as scheduled and opted to continue receiving OL study treatment continued to receive macitentan 10mg in OLE period.
Period: Double-blind (DB) Treatment Period
Arm/Group | Macitentan 10 mg | Placebo
Started | 43 | 42
Completed | 39 | 41
Not Completed | 4 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Open-label (OL) Treatment Period
Arm/Group | Macitentan 10 mg | Placebo
Started | 80 | 0
Completed | 71 | 0
Not Completed | 9 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 4 | 0
Period: OL Extension Period
Arm/Group | Macitentan 10 mg | Placebo
Started | 33 (Participants(French site) who completed DB,OL periods, consented receiving macitentan in OLE period.) | 0
Completed | 27 | 0
Not Completed | 6 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Macitentan 10 mg: Participants received Macitentan 10 milligram (mg) film-coated tablets orally once daily for 12 weeks in Double-blind treatment period.
- Placebo: Participants received Macitentan matching placebo film-coated tablets orally once daily for 12 weeks in Double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Macitentan 10 mg | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 29 | 64
  >=65 years | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (8.7) | 59.0 (9.5) | 58.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 22 | 22 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 19 | 15 | 34
  Unknown or Not Reported | 18 | 21 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 23 | 21 | 44
  Other | 1 | 0 | 1
  Not Applicable | 18 | 21 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23
  Brazil | 2 | 3 | 5
  Czech Republic | 1 | 3 | 4
  France | 18 | 21 | 39
  Germany | 4 | 4 | 8
  Spain | 4 | 0 | 4
  United Kingdom | 2 | 0 | 2
Pulmonary arterial hypertension (PAH)-specific therapy [Count of Participants; unit: Participants] — As per randomization stratification, 63.5% of patients were receiving a pulmonary arterial hypertension (PAH)-specific therapy at baseline.
  Participants
    Yes | 27 | 27 | 54
    No | 16 | 15 | 31
Body Mass Index (BMI) at baseline [Mean (Standard Deviation); unit: Kilogram per meter^2 (Kg/m^2)] | 29.01 (4.79) | 29.33 (4.04) | 29.17 (4.41)
Time since portal hypertension diagnosis [Median (Inter-Quartile Range); unit: Months] | 23 [5 to 80] | 31 [4 to 69] | 25 [7 to 76]
Time since PAH diagnosis [Median (Inter-Quartile Range); unit: Months] | 7 [2 to 33] | 12 [1 to 37] | 10 [2 to 36]
Pulmonary vascular resistance (PVR) at baseline (calculated) [Mean (Standard Deviation); unit: Dyn*sec/cm^5] | 552.4 (192.8) | 521.7 (163.3) | 537.2 (178.4)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline to Week 12 in Pulmonary Vascular Resistance (PVR).
Description: The relative change from baseline to Week 12 in PVR is expressed as a ratio of Week 12 to baseline PVR.
Time Frame: From enrollment/baseline to Week 12 in the Double Blind (DB) treatment period
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
ratio | 0.63 [0.58 to 0.67] | 0.98 [0.91 to 1.05]
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; The null hypothesis (change of PVR at Week 12 as a ratio of baseline PVR in subjects treated with placebo or macitentan is the same) is tested on the primary endpoint by means of an analysis of covariance (ANCOVA) model on the log(e) transformed ratio of PVR at Week 12 to baseline PVR; Test type: Superiority; p = 0.0001, ANCOVA; ANCOVA model adjusted by treatment, background PAH-specific therapy at baseline and region as factors & log-transformed PVR at baseline as a covariate; ratio of geometric means = 0.65, 95% CI 2-sided [0.59 to 0.72]

2. Secondary Outcome: Change From Baseline to Week 12 in 6-minute Walk Distance (6MWD)
Description: The purpose of the six minute walk is to test exercise tolerance and capacity. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
meter
  6MWD at baseline | 385.8 (99.97) | 383.2 (108.90)
  6MWD at Week 12 | 392.2 (98.46) | 380.8 (114.98)
  Change of 6MWD from baseline to Week 12 | 6.4 (65.74) | -2.4 (43.65)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; The main analysis on 6MWD was performed using a mixed-effect model repeated measure (MMRM) adjusted for treatment, visit, region, PAH-specific therapy at baseline, and treatment-by-visit interaction as factors, and baseline 6MWD and WHO functional class (FC) as covariates; Test type: Superiority; p = 0.4264, mixed-effect model repeated measure — No adjustment was made for multiplicity for secondary endpoints, therefore all corresponding p-values provided are of an exploratory nature; Least squares (LS) mean difference = 9.73, 95% CI 2-sided [-14.50 to 33.95] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in 6MWD (LS mean difference macitentan 10 mg - placebo)

3. Secondary Outcome: Change From Baseline to Week 12 in WHO Functional Class (FC)
Description: Changes from baseline to Week 12 in WHO FC were dichotomized as worsening (i.e., change > 0) versus no change or improvement (i.e., change ≤ 0). Class I: no symptoms with exercise or at rest. No limitation of activity. Class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing a flight of stairs, grocery shopping, or making the bed). Class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. Class IV: symptoms at rest (e.g. dyspnea and/or fatigue) and inability to carry out any physical activity without symptoms. Patients in class IV manifest signs of right heart failure.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
Participants
  WHO FC I at baseline | 1 | 1
  WHO FC II at baseline | 27 | 23
  WHO FC III at baseline | 15 | 18
  WHO FC IV at baseline | 0 | 0
  WHO FC I at Week 12 | 3 | 4
  WHO FC II at Week 12 | 27 | 23
  WHO FC III at Week 12 | 13 | 15
  WHO FC IV at Week 12 | 0 | 0
  Improved from baseline to Week 12 | 9 | 7
  Worsened from baseline to Week 12 | 6 | 1
  Unchanged from baseline to Week 12 | 28 | 34
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; A logistic regression model (exact) adjusted for treatment, PAH-specific therapy at baseline, and region as covariates was used to analyze worsening in WHO FC; Test type: Superiority; p = 0.1278, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 6.253, 95% CI 2-sided [0.714 to 298.376]

4. Secondary Outcome: Change From Baseline to Week 12 in the Biomarker N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP functions as a strong indicator of prognosis in patients with pulmonary hypertension (PH). The relative change from baseline to Week 12 in NT-proBNP is expressed as a ratio of Week 12 to baseline NT-proBNP.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Population: Full Analysis Set(FAS): All randomized participants who received at least one dose of study drug in DB treatment, have baseline value for PVR, evaluated As per assigned treatment. Here, 'N'(number of participants analyzed included population included participants with available baseline data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 41 | 40
ratio | 0.86 [0.67 to 1.11] | 1.04 [0.81 to 1.34]
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.3951, ANCOVA — [p-value comment as in outcome 2, analysis 1]; ratio of geometric means = 0.874, 95% CI 2-sided [0.639 to 1.196]

5. Secondary Outcome: Change From Baseline to Week 12 in Mean Right Atrial Pressure (mRAP)
Description: mRAP is the mean blood pressure in the right atrium of the heart.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 42 | 42
mmHg
  mRAP at baseline | 7.3 (3.74) | 6.7 (3.60)
  mRAP at Week 12 | 9.0 (5.32) | 7.0 (2.93)
  Change in mRAP from baseline to Week 12 | 1.6 (5.55) | 0.3 (3.29)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.0637, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares (LS) mean difference = 1.67, 95% CI 2-sided [-0.10 to 3.44] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in mRAP (LS mean difference macitentan 10 mg - placebo)

6. Secondary Outcome: Change From Baseline to Week 12 in Mean Pulmonary Artery Pressure (mPAP)
Description: mPAP is the mean blood pressure inside the pulmonary artery which moves the blood from the heart to the lungs. Monitoring of mPAP can detect small changes in the function of the heart.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
mmHg
  mPAP at baseline | 46.4 (7.89) | 43.8 (8.52)
  mPAP at Week 12 | 40.0 (7.61) | 44.2 (8.26)
  Change in mPAP at Week 12 | -6.4 (4.94) | 0.4 (7.04)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares (LS) mean difference = -5.99, 95% CI 2-sided [-8.40 to -3.57] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in mPAP (LS mean difference macitentan 10 mg - placebo)

7. Secondary Outcome: Change From Baseline to Week 12 in Cardiac Index
Description: The cardiac index is an assessment of the function of the heart and relates the cardiac output to the patient's body size (the patient's body surface area).
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
L/min/m^2
  Cardiac index at baseline | 3.1 (0.83) | 2.9 (0.76)
  Cardiac index at Week 12 | 3.7 (1.04) | 3.0 (0.82)
  Change in cardiac index at Week 12 | 0.6 (0.8) | 0.1 (0.6)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.0009, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares (LS) mean difference = 0.52, 95% CI 2-sided [0.22 to 0.81] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in cardiac index (LS mean difference macitentan 10 mg - placebo)

8. Secondary Outcome: Change From Baseline to Week 12 in Total Pulmonary Resistance (TPR)
Description: TPR is the resistance the pulmonary circulation that must be overcome in order for the blood flow to occur. It takes into account the blood pressure in the pulmonary arteries and the cardiac output. It is an important measurement to monitor the function of the pulmonary circulation and detect disease progression or improvement.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Measure: Mean (Standard Deviation); unit: dyn*sec/cm^5
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 43 | 42
dyn*sec/cm^5
  TPR at baseline | 689.3 (228.59) | 671.5 (199.73)
  TPR at Week 12 | 489.4 (157.13) | 653.1 (197.88)
  Change in TPR from baseline to Week 12 | -199.8 (163.06) | -18.3 (135.28)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares (LS) mean difference = -171.48, 95% CI 2-sided [-223.67 to -119.30] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in TPR (LS mean difference macitentan 10 mg - placebo)

9. Secondary Outcome: Change From Baseline to Week 12 in Mixed Venous Oxygen Saturation (SVO2)
Description: SVO2 help assess tissue oxygen delivery. It describes the percentage of oxygen bound to hemoglobin in the blood which returns to the heart. This reflects the amount of residual oxygen in the blood after oxygen extraction by the tissues throughout the body.
Time Frame: From enrollment/baseline to Week 12 in the DB treatment period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent of oxygen bound to hemoglobin
Arm/Group | Macitentan 10 mg | Placebo
Number analyzed (Participants) | 41 | 41
percent of oxygen bound to hemoglobin
  SVO2 at baseline | 69.2 (9.87) | 69.9 (5.34)
  SVO2 at Week 12 | 70.3 (7.07) | 70.7 (8.58)
  Change in SVO2 from baseline to Week 12 | 1.1 (6.70) | 0.8 (7.81)
Statistical Analysis 1: Comparison: Macitentan 10 mg vs Placebo; Test type: Superiority; p = 0.9844, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares (LS) mean difference = 0.03, 95% CI 2-sided [-2.85 to 2.91] — The estimated value refers to a between-treatment analysis of change from baseline to Week 12 in SVO2 (LS mean difference macitentan 10 mg - placebo)

ADVERSE EVENTS:
Time Frame: Up to 3.4 years
Description: The Safety Set (SS) included all participants who received at least one dose of study treatment.
Groups:
- Double-Blind (DB) Period: Macitentan 10 mg: Participants received Macitentan 10 milligram (mg) film-coated tablets orally once daily for 12 weeks during DB treatment period.
- DB Period: Placebo: Participants received Macitentan matching placebo film-coated tablets orally once daily for 12 weeks during DB treatment period.
- Open-Label (OL) Period: Macitentan 10 mg: Participants received Macitentan 10 milligram (mg) film-coated tablets orally once daily for 12 weeks in Double-blind treatment period. Participants who completed DB treatment period continued to receive macitentan 10 mg for 12 weeks (up to Week 24) in OL treatment period.
- OL Extension Period: Macitentan 10 mg: Participants received Macitentan 10 milligram (mg) film-coated tablets orally once daily for 12 weeks in Double-blind treatment period. Participants who completed DB treatment period continued to receive macitentan 10 mg for 12 weeks (up to Week 24) in OL treatment period . Participants (who were randomized at French sites) who completed the core phase of the study as scheduled and opted to continue receiving OL study treatment continued to receive macitentan 10 mg in OLE period.
Arm/Group | Double-Blind (DB) Period: Macitentan 10 mg | DB Period: Placebo | Open-Label (OL) Period: Macitentan 10 mg | OL Extension Period: Macitentan 10 mg
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 4/80 | 2/33
Serious Adverse Events (participants affected / at risk) | 9/43 | 6/42 | 18/80 | 11/33
Other Adverse Events (participants affected / at risk) | 34/43 | 32/42 | 62/80 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind (DB) Period: Macitentan 10 mg (N=43) | DB Period: Placebo (N=42) | Open-Label (OL) Period: Macitentan 10 mg (N=80) | OL Extension Period: Macitentan 10 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 2 | 1 | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Duodenal Vascular Ectasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Escherichia Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Liver Function Test Increased (Investigations) | 0 | 0 | 1 | 0
Troponin I Increased (Investigations) | 1 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 1 | 0 | 0
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aneurysm Repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind (DB) Period: Macitentan 10 mg (N=43) | DB Period: Placebo (N=42) | Open-Label (OL) Period: Macitentan 10 mg (N=80) | OL Extension Period: Macitentan 10 mg (N=33)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 9 | 5
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 1
Conjunctival Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Diabetic Retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 2 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1
Eye Oedema (Eye disorders) | 0 | 0 | 0 | 1
Eye Pruritus (Eye disorders) | 1 | 0 | 0 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 1 | 0
Meibomian Gland Dysfunction (Eye disorders) | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anal Polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Duodenal Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Portal Hypertensive Gastropathy (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Varices Oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 1 | 4 | 3
Chest Pain (General disorders) | 0 | 1 | 1 | 1
Face Oedema (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0
Generalised Oedema (General disorders) | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 3 | 2
Localised Oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 10 | 5 | 13 | 5
Pain (General disorders) | 0 | 1 | 1 | 0
Peripheral Swelling (General disorders) | 2 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0
Temperature Intolerance (General disorders) | 0 | 0 | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic Mass (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 3 | 13
Candida Infection (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 2
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 4 | 7
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 2
Sinusitis Fungal (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 1 | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ammonia Increased (Investigations) | 1 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0
Blood Potassium Decreased (Investigations) | 1 | 0 | 1 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 1 | 0
Blood Sodium Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 0 | 1 | 0
Blood Urine Present (Investigations) | 1 | 0 | 0 | 0
Brain Natriuretic Peptide Increased (Investigations) | 0 | 0 | 1 | 0
Coronavirus Test Positive (Investigations) | 0 | 0 | 1 | 0
Haematocrit Decreased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 3 | 0 | 3 | 0
Intestinal Transit Time Decreased (Investigations) | 1 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 0
Total Bile Acids Increased (Investigations) | 1 | 0 | 1 | 0
Urine Output Decreased (Investigations) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Folate Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Magnesium Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sebaceous Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 5 | 1
Headache (Nervous system disorders) | 7 | 7 | 10 | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol Abuse (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 5
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Bendopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Portopulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Umbilical Haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alcohol Use (Social circumstances) | 0 | 0 | 0 | 1
Inguinal Hernia Repair (Surgical and medical procedures) | 0 | 0 | 0 | 1
Oesophageal Variceal Ligation (Surgical and medical procedures) | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 3 | 0
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation Decreased (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Groin Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intestinal Transit Time Abnormal (Investigations) | 0 | 1 | 0 | 0
Venous Pressure Jugular Increased (Investigations) | 0 | 1 | 0 | 0
Weight Increased (Investigations) | 0 | 1 | 0 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Injection (Surgical and medical procedures) | 0 | 1 | 0 | 0
Skin Neoplasm Excision (Surgical and medical procedures) | 0 | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02382016/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT02382016/SAP_002.pdf